CLINICAL TRIAL: NCT05711329
Title: The Aim of This Study is to Determine the Accuracy of the Self-reported Parameters (Compared to Measurement Performed by the Physician) and the Influence of OSA Screening Scores.
Brief Title: Comparison of Methodology Proposed by the SFAR for the Detection by Videoconference of Obstructive Sleep Apnea.
Status: Not yet recruiting | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, FAACD, Head of Department, Astes
Other Study IDs: Visio-PSG
Record Dates: First submitted 2023-01-24; First posted 2023-02-03 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Patients in this group will serve to validate the accuracy of the French method to detect OSA patients in comparison with PSG results.
  Interventions: Other: Accuracy

INTERVENTIONS:
Other: Accuracy — We will validate the accuracy of the method proposed by the SFAR to detect OSA patients via videoconference (in comparison with the results of the PSG).

SUMMARY:
The SFAR (French society of anesthesiology and ICU) proposed a method to detect OSA (Obstructive Sleep Apnea) patients via videoconference. The aim of this study is to compare the result of this method with the results of polysomnography (PSG) which remains the gold standard in the detection of OSA patients.

DETAILED DESCRIPTION:
The SFAR (French society of anesthesiology and ICU) proposed a method to detect OSA (Obstructive Sleep Apnea) patients via videoconference. The aim of this study is to compare the result of this method with the results of polysomnography (PSG) which remains the gold standard in the detection of OSA patients.

Other methods, such as a predictive score, also exist. The accuracy of the French method compared to PSG and the predictive scores is to be determined.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in the Clinique Saint-Luc of Bouge for a polysomnography

Exclusion Criteria:

* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population to validate the method proposed by the SFAR to detect OSA patients via videoconference.
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation of the method proposed by the SFAR by comparison with results of polysomnography. | 1 month
  Validation (or not) of the method proposed by the SFAR to detect OSA patient va videoconference.
  The SFAR proposed a method to detect OSA patients throughout a videoconference. This method consists in requesting the patient to go around his neck with his two hands. However, this method has not been validated. The outcome of the study is to validate or invalidate the method proposed by the SFAR in comparison with the results of polysomnography (which remains the gold standard for the diagnosis of OSA patients).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, MD, PhD, Principal Investigator — Astes

IPD SHARING:
Plan to Share IPD: No